CLINICAL TRIAL: NCT07065734
Title: NEgative prEssure Wound Therapy in Renal Transplant - NEWER Trial
Brief Title: NEgative prEssure Wound Therapy in Renal Transplant
Acronym: NEWER
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centro Hospitalar De São João, E.P.E. (Other)
Collaborators: Universidade do Porto (Other)
Responsible Party: Principal Investigator, Alberto Costa Silva, Principal Investigator, Centro Hospitalar De São João, E.P.E.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 351-2022
Record Dates: First submitted 2025-06-23; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Transplant Complication; Renal Transplant; Wound Complication
Keywords: transplant complication; renal transplant; wound complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NPWT group (Active Comparator): Patients who received negative pressure wound therapy
  Interventions: Device: NWPT group
- Standard group (No Intervention): Patients who received standard dressing

INTERVENTIONS:
Device: NWPT group — Patients submitted to negative pressure wound therapy
  Arms: NPWT group

SUMMARY:
This is a prospective study involving patients undergoing open renal transplant. Renal transplant recipients were randomly divided into two groups: the NPWT group, which received NPWT, and the Standard group, which received standard wound dressings.

DETAILED DESCRIPTION:
This is a prospective study involving patients undergoing open renal transplant between January 2023 and August 2024. Pediatric patients, those requiring surgical reinterventions within the first 3 postoperative months, and patients allergic to NPWT components were excluded from the study. Renal transplant recipients were randomly divided into two groups: the NPWT group, which received NPWT, and the Standard group, which received standard wound dressings. NPWT (PICO by Smith & Nephew) was applied intraoperatively at 80 mmHg and maintained for 7 days. Wound evaluations were performed at 7, 14, 30, and 90 days post-operatively. If dehiscence was present, it was classified as either deep or superficial based on the involvement of the aponeurosis. Patients were assessed for wound infection using the ASEPSIS score, pain with a visual analogue scale, and quality of life using the EQ-5D questionnaire. Scar healing was also evaluated at 30 and 90 days post-operatively with the POSAS score

ELIGIBILITY:
Inclusion Criteria:

* All patients submitted to kidney transplant

Exclusion Criteria:

* Pediatric patients, those requiring surgical reinterventions within the first 90 days postoperative, patients allergic to NPWT components, orthotopic transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Wound dehiscence | First 90 days after surgery
  Wound dehiscence - superficial or deep

SECONDARY OUTCOMES:
Wound infection | First 90 days after surgery
  ASEPSIS score - (Additional treatment, Serous discharge, Erythema, Purulen exudates, Separation of deep tissues, Isolation of bacteria, Stay in hospital score); 0-10 points; higher score = worse outcome
Pain associated with incision | First 90 days after surgery
  Visual analogue scale; score 0-10; higher score=worse outcome
Quality of life associated with incision | First 90 days after surgery
  EQ-5D questionnaire (The 5-level quality of life version 5); score 0 -100 ; highest score=better outcome
Scar healing | First 90 days after surgery
  POSAS score (The Patient and Observer Scar Assessment Scale); score 1-10; highest score=worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: João Alturas Silva, PhD, Study Director — São João University Hospital
Locations (1):
- São João University Hospital, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared upon reasonable request after consideration from local Ethics Comission

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-10): https://cdn.clinicaltrials.gov/large-docs/34/NCT07065734/Prot_SAP_000.pdf